CLINICAL TRIAL: NCT06662760
Title: A Phase I Clinical Study of TQB3002 in Patients With Advanced Cancers
Brief Title: Clinical Trial of TQB3002 in Patients With Advanced Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB3002-I-01
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-09

CONDITIONS: Advanced Cancer

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TQB3002 Tablets (Experimental): TQB3002 Tablets, 28 days as a treatment cycle
  Interventions: Drug: TQB3002 Tablets

INTERVENTIONS:
Drug: TQB3002 Tablets — TQB3002 is a fourth-generation small molecule Epidermal growth factor receptor (EGFR) inhibitor, which inhibits relevant tyrosine kinase activity and intracellular phosphorylation process by competitively binding to Adenosine triphosphate (ATP) site of intracellular tyrosine kinase binding domain, thereby inhibiting EGFR downstream signaling, ultimately achieving the purpose of inhibiting tumor growth.

SUMMARY:
This is a Phase I study to evaluate the safety, tolerability, and efficacy of TQB3002 in subjects with advanced cancers

ELIGIBILITY:
Inclusion Criteria:

* Subjects voluntarily joined this study, signed the informed consent form, and had good compliance；
* Age: ≥ 18 years old; Eastern Cooperative Oncology Group (ECOG) score: 0-1 ; Expected survival of more than 3 months；
* Histologically or cytologically diagnosed with advanced cancers
* Subjects with advanced malignancies who have failed standard therapy or lack effective treatment
* Major organs are functioning well；
* Female and male subjects of childbearing potential should agree to practice contraception for the duration of the study and for 6 months after the end of the study.

Exclusion Criteria:

* Current concomitant presence of other malignancies within 5 years prior to the first dose；
* Unresolved toxicity above CTCAE Grade 1 due to any prior anti-tumor therapy
* Significant surgical treatment, biopsy, or significant traumatic injury within 4 weeks prior to the first dose
* Long-term unhealed wounds or fractures
* Cerebrovascular accident (including transient ischemic attack, intracerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism within 6 months prior to the first dose
* Swallowing dysfunction, active gastrointestinal diseases or other diseases that significantly affect the absorption, distribution, metabolism and excretion of the study drug, or previous subtotal gastrectomy
* A history of psychotropic drug abuse and cannot be abstained from or have a mental disorder
* Subjects with any severe and/or uncontrolled disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-12-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | During the first 28 days
  DLT will be defined as toxicities that meet pre-defined severity criteria(according to the NCI CTCAE v5.0 toxicity assessment criteria), and assessed as having a suspected relationship to study drug that occurred within the first cycle(28days) of treatment.
Maximum tolerated dose (MTD) | During the first 28 days
  MTD is defined as the highest dose at which dose-limiting toxicity (DLT) occurred in less than 33% of patients.

SECONDARY OUTCOMES:
Half-life (T1/2) | Before administration (-1 hour ~ 0 hour), 0.5, 1, 2, 3, 4, 6, 8h , 12, 24, 48, 72, 96 and 168 hours after administration
  Terminal half-life (T1/2)
The area under the curve (AUC) | Before administration (-1 hour ~ 0 hour), 0.5, 1, 2, 3, 4, 6, 8h , 12, 24, 48, 72, 96 and 168 hours after administration
  The area under the curve (AUC) of serum concentration of TQB3002
Apparent Plasma Clearance (CL) | Before administration (-1 hour ~ 0 hour), 0.5, 1, 2, 3, 4, 6, 8h , 12, 24, 48, 72, 96 and 168 hours after administration
  Apparent plasma clearance of TQB3002
Apparent volume of distribution (Vz) | Before administration (-1 hour ~ 0 hour), 0.5, 1, 2, 3, 4, 6, 8h , 12, 24, 48, 72, 96 and 168 hours after administration
  The ratio of the amount of TQB3002 in the body to the blood concentration
Minimum concentration (Cmin) | Before administration (-1 hour ~ 0 hour), 0.5, 1, 2, 3, 4, 6, 8h , 12, 24, 48, 72, 96 and 168 hours after administration
  Minimum observed concentration (Cmin) of TQB3002

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Nanchang University, Nanchang, Jiangxi
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi’an, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Mianyang Central Hospital, Mianyang, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan